CLINICAL TRIAL: NCT04975620
Title: Comparison of Two Types of Biopsy Needles for Endoscopic Ultrasound-guided Fine Needle Biopsy (EUS-FNB) in Solid Pancreatobiliary Mass Lesions
Brief Title: Comparison of Two Types of Biopsy Needles for EUS-FNB in Solid Pancreatobiliary Mass Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Mehdi Mohamadnejad, Associate professor of medicine, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IR.TUMS.DDRI.REC.1400.008
Record Dates: First submitted 2021-07-04; First posted 2021-07-23 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Neoplasms
Keywords: Fine needle biopsy; Endoscopic ultrasonography; Diagnosis
MeSH Terms: conditions — Pancreatic Neoplasms; Disease | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The pathologists who assess the FNB specimens are blinded on the needle type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Franseen needle with three symmetric cutting edges (Experimental): These patients will undergo endoscopic ultrasound-guided fine needle biopsy using the Franseen needle (Acquire FNB needle; Boston Scientific): eight back and forth movements within the lesion will be performed with simultaneous minimal negative pressure provided by withdrawing the needle stylet slowly. Four passes of FNB will be made from each mass lesion and the specimens from each pass will be placed in different containers for cell block preparation and histologic evaluation.
  Interventions: Device: Fine needle biopsy
- Multi-blade needle with three-prong tip with one tip longer than the other two (Experimental): These patients will undergo endoscopic ultrasound-guided fine needle biopsy using a multi-blade three-prong tip needle (Trident; Microtech): eight back and forth movements within the lesion will be performed with simultaneous minimal negative pressure provided by withdrawing the needle stylet slowly. Four passes of FNB will be made from each mass lesion and the specimens from each pass will be placed in different containers for cell block preparation and histologic evaluation.
  Interventions: Device: Fine needle biopsy

INTERVENTIONS:
Device: Fine needle biopsy — Taking biopsy from solid pancreatobiliary mass lesions with 8 back and forth movement of the needle within the lesion with slow withdrawal of the stylet

SUMMARY:
EUS-guided tissue acquisition is an established modality to diagnose malignancies of the pancreas and extrahepatic bile ducts. In the recent years fine needle biopsy (FNB) needles have largely replaced fine needle aspiration (FNA) for EUS-guided tissue acquisition. The Acquire FNB needle is a Franseen needle which has three symmetric cutting edges to obtain core tissue specimens. The Trident FNB needle has been recently introduced to the market for EUS-guided tissue acquisition. It has a multi-blade three-prong tip which one of the tips is longer than the other two.

The aim of this study is to prospectively compare these two types of needle in term of diagnostic accuracy, and safety profile.

DETAILED DESCRIPTION:
Patients with solid mass lesions in the pancreas or extrahepatic biliary system will be randomly assigned to one of two types of FNB needle. Four passes of FNB will be acquired from the mass lesion in each patient. The primary aim is to compare sensitivity of two types of FNB needle to diagnose malignancy. Also, each pass of FNB needle will be assessed separately by two expert pathologists to determine per-pass sensitivity of two types of FNB needles.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients 18 years of age or older with solid mass lesions in the pancreas or extrahepatic biliary system

Exclusion Criteria:

* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Decline to participate in the study and sign the informed consent form
* Cystic lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of EUS-FNB sensitivity using two types of FNB needles | 6 months
  Comparison of EUS-FNB sensitivity using two types of FNB needles

SECONDARY OUTCOMES:
Comparing per-pass sensitivity in two types of FNB needles | 6 months
  Comparing per-pass sensitivity in two types of FNB needles
Comparing the adequacy of specimen for each pass in two types of FNB needles | 6 months
  Comparing the adequacy of specimen for each pass in two types of FNB needles
Comparing the rate of core tissue acquisition for each pass in two types of FNB needles | 6 months
  Comparing the rate of core tissue acquisition for each pass in two types of FNB needles
Comparing specimen cellularity for each pass in two types of FNB needles | 6 months
  Comparing specimen cellularity for each pass in two types of FNB needles
Comparing the score of blood content n for each pass in two types of FNB needles. | 6 months
  Comparing the score of blood content n for each pass in two types of FNB needles. (The blood content is scored from 1 to 3 in which 1 represents minimal presence of blood in the specimen).

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Diseases Research Institute, Shariati Hospital, North Kargar Ave.,, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mohamadnejad M, Mullady D, Early DS, Collins B, Marshall C, Sams S, Yen R, Rizeq M, Romanas M, Nawaz S, Ulusarac O, Hollander T, Wilson RH, Simon VC, Kushnir V, Amateau SK, Brauer BC, Gaddam S, Azar RR, Komanduri S, Shah R, Das A, Edmundowicz S, Muthusamy VR, Rastogi A, Wani S. Increasing Number of Passes Beyond 4 Does Not Increase Sensitivity of Detection of Pancreatic Malignancy by Endoscopic Ultrasound-Guided Fine-Needle Aspiration. Clin Gastroenterol Hepatol. 2017 Jul;15(7):1071-1078.e2. doi: 10.1016/j.cgh.2016.12.018. Epub 2016 Dec 23. PMID 28025154
- [Result] Sadeghi A, Mohamadnejad M, Islami F, Keshtkar A, Biglari M, Malekzadeh R, Eloubeidi MA. Diagnostic yield of EUS-guided FNA for malignant biliary stricture: a systematic review and meta-analysis. Gastrointest Endosc. 2016 Feb;83(2):290-8.e1. doi: 10.1016/j.gie.2015.09.024. Epub 2015 Sep 28. PMID 26422979
- [Result] Bang JY, Hebert-Magee S, Navaneethan U, Hasan MK, Hawes R, Varadarajulu S. EUS-guided fine needle biopsy of pancreatic masses can yield true histology. Gut. 2018 Dec;67(12):2081-2084. doi: 10.1136/gutjnl-2017-315154. Epub 2017 Oct 7. No abstract available. PMID 28988195
- [Derived] Mohamadnejad M, Mirzaie V, Sotoudeh M, Nikmanesh A, Hosseini R, Muthusamy R. Comparing per-pass performance of 2 types of needles for EUS-guided fine-needle biopsy sampling of pancreatobiliary masses in a randomized trial. Gastrointest Endosc. 2023 Sep;98(3):371-380. doi: 10.1016/j.gie.2023.04.2070. Epub 2023 Apr 23. PMID 37098399